CLINICAL TRIAL: NCT04579848
Title: The Methotrexate in ERosive INflammatory Osteoarthritis (MERINO) Trial: A Randomized Placebo-controlled Trial to Investigate Clinical Efficacy and Safety of Methotrexate in Erosive Inflammatory Hand Osteoarthritis.
Brief Title: Methotrexate in Erosive Inflammatory Hand Osteoarthritis
Acronym: MERINO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ida Kristin Haugen, Senior researcher, doctor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIA2020-01
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hand Osteoarthritis; Erosive Osteoarthritis
MeSH Terms: interventions — Methotrexate; Folic Acid

STUDY DESIGN:
Intervention Model Description: An investigator-initiated, randomized, double-blinded, placebo-controlled, parallel-group, single-center, phase IV, superiority study, exploring the effect of methotrexate on pain, function and structural outcomes in erosive inflammatory hand osteoarthritis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical placebo cannot be produced due to text, color and shape of methotrexate tablets. Thus, both placebo and methotrexate will be encapsulated to ensure blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methotrexate (Active Comparator): Methotrexate oral x 1/week; weekly starting dose 15 mg for two weeks, followed by 20 mg the remaining weeks.
  Additional Folic acid 1mg prescribed daily.
  Interventions: Drug: Methotrexate Tablets; Drug: Folic Acid 1 MG
- Placebo (Placebo Comparator): 3 capsules per week for two weeks, followed by 4 capsules the remaining weeks.
  Additional Folic acid 1mg prescribed daily.
  Interventions: Drug: Placebo; Drug: Folic Acid 1 MG

INTERVENTIONS:
Drug: Methotrexate Tablets — Methotrexate 2.5mg oral tablet.
  Arms: Methotrexate
Drug: Placebo — Placebo capsule
  Arms: Placebo
Drug: Folic Acid 1 MG — Folic acid

SUMMARY:
A placebo-controlled randomized controlled trial exploring the effect of methotrexate on pain, function and structural outcomes in erosive inflammatory hand osteoarthritis.

DETAILED DESCRIPTION:
The trial will include Norwegian adult males and females with symptomatic erosive inflammatory hand osteoarthritis.

Participants will be randomized 1:1 to either:

1. Methotrexate oral x 1/week; weekly starting dose 15 mg for two weeks, followed by 20 mg the remaining weeks (intervention group). Dosage can be reduced to as low as 10 mg if higher doses are not tolerated.
2. Placebo (control group).

Both arms will receive folic acid 1mg daily.

The treatment duration for both groups is 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Finger joint pain 40-80 on 0-100 visual analog scale (VAS) with insufficient pain relief from, inability to tolerate or contra-indications to oral paracetamol and/or NSAIDs, and hand symptoms (pain, aching, or stiffness) on most days the previous 6 weeks before randomization.
* Hand OA according to the American College of Rheumatology (ACR) criteria, at least 1 distal (DIP) or proximal interphalangeal (PIP) joint of the 2nd-5th finger with radiographic pre-erosive (J-phase) or erosive disease (E-phase) according to the Verbruggen-Veys anatomical phase system, and at least two DIP/PIP joints with power Doppler signal of at least grade 1 or grey-scale synovitis of at least grade 2 on ultrasound.

Exclusion Criteria:

A full list of the exclusion criteria for this study comprised the following:

* Contraindications to methotrexate:

  * Abnormal renal function, defined as serum creatinine >142 µmol/L in women and >168 µmol/L in men, or a glomeruli filtration rate (GFR) <40 mL/min/1.73 m2.
  * Abnormal liver function, defined as transaminases above the upper normal limit, active or previous hepatitis B or C infection, or known cirrhosis
  * Lung fibrosis (maximum 6 months old x-ray), active infection, or reduced hematopoiesis (i.e. anemia, leukopenia and/or thrombocytopenia).
  * Planned pregnancy within 18 months after screening (men/women), and pregnancy, breastfeeding, or insufficient anti-conception therapy for female fertile participants. Contraception should be maintained during treatment and until the end of systemic exposure, i.e. 3 months after methotrexate discontinuation. Sufficient anti-conception therapy consists of intra-uterine device (coil) or hormonal anti-conception (birth control pills, implant, intra-uterine system, dermal patch, vaginal ring, or injections).
  * Alcohol or other drug abuse in the last year.
  * Intolerance to lactose.
* Chronic inflammatory rheumatic diseases (such as rheumatoid arthritis and psoriatic arthritis or gout), active inflammatory bowel disease, or positive rheumatoid factor or anti-CCP antibodies.
* Other severe co-morbidities such as hemochromatosis, fibromyalgia, psoriasis, blood dyscrasias, and coagulation disorders, history of malignancy (except successfully treated squamous or basal cell skin carcinoma), uncontrolled diabetes mellitus, severe hypertension, unstable ischemic heart disease, severe heart failure, severe pulmonary disease, severe and/or opportunistic infections and/or chronic infections, active tuberculosis, positive human immunodeficiency virus (HIV) status, recent stroke, bone marrow hypoplasia, or demyelinating diseases of the central nervous system.
* Other likely causes of hand symptoms: thoracic outlet syndrome, carpal tunnel disease, diabetic cheiropathy, injury in finger joints previous 6 months, or palmar tenosynovitis/trigger finger.
* Oral or intra-muscular steroids in the previous month
* Intra-articular treatments or aspirations of any kind of any joint in the hands 3 months before inclusion
* Analgesics or NSAIDs, unless stable dosage for ≥1 month.
* Symptomatic slow-acting drugs for OA (SYSADOA), unless stable dose for ≥3 months and require stable dose throughout the study.
* Disease-modifying osteoarthritis drugs (DMOADs) previous three months.
* Scheduled hand surgery during study participation.
* Planning to start other treatments for hand OA in the study participation period.
* Not able to adhere to the study visit schedule and protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Finger pain on a visual analogue scale | 6 months
  Difference in self-reported finger joint pain previous 48 hours on a 0-100 mm scale at 6 months of treatment; higher value indicate worse outcome.

SECONDARY OUTCOMES:
Finger pain on a visual analogue scale | Month 1, 3, 9 and 12.
  Self-reported finger pain previous 48 hours on a 0-100 mm scale; higher value indicate worse outcome.
Thumb pain on a visual analogue scale | Month 1, 3, 6, 9 and 12.
  Self-reported thumb pain previous 48 hours on a 0-100 mm scale; higher value indicate worse outcome.
Pain most painful finger joint on a visual analogue scale | Month 1, 3, 6, 9 and 12.
  Pain most painful finger joint last 48 hours on a 0-100 mm scale; higher value indicate worse outcome.
Patient-reported disease activity on a visual analogue scale | Month 1, 3, 6, 9 and 12.
  Patient-reported disease activity last 48 hours on a 0-100 mm scale; higher value indicate worse outcome.
Pain all joints on a visual analogue scale | Month 1, 3, 6, 9 and 12.
  Pain all joints last 48 hours on a 0-100 mm scale; higher value indicate worse outcome.
Hand diagram pain | Month 6.
  Finger pain and thumb base pain (yes/no) on hand diagram
Body diagram pain | Month 6.
  Pain in other joints (yes/no) on body diagram
AUSCAN | Month 1, 3, 6, 9 and 12.
  Australian/Canadian hand index (AUSCAN), sum score 0-60, higher value indicate worse outcome.
OMERACT-OARSI responder criteria | Month 1, 3, 6, 9 and 12.
  Fulfillment of Outcome Measures in Rheumatology Osteoarthritis Research Society International (OMERACT-OARSI) responder criteria.
EQ-5D | Month 1, 3, 6, 9 and 12.
  Quality-adjusted life years (QALYs) based on the health-related utility scores measured by the generic instrument EuroQol 5 dimensions (EQ-5D), sum score 5-35, higher value indicate worse outcome, in addition to a 0-100 visual analogue scale where higher value indicate better outcome.
MHOQ | Month 6.
  Michigan Hand Outcomes Questionnaire (MHOQ) pain and physical function subscales; function subscale range 10-50, higher value indicate worse outcome; task subscale range 17-85, higher value indicate worse outcome; work subscale range 5-25, higher value indicate worse outcome; pain subscale range 10-48, higher value indicate better outcome.
Grip strength | Month 1, 3, 6, 9 and 12.
  Grip strength (in kg; using a hand dynamometer)
HOOS-12 | Month 6.
  Hip disability and Osteoarthritis Outcome Score (HOOS)-12, range 12-60, higher value indicate worse outcome.
KOOS-12 | Month 6.
  Knee injury and Osteoarthritis Outcome Score (KOOS)-12, range 12-60, higher value indicate worse outcome.
Concomitant medication | Month 1, 3, 6, 9 and 12.
  Concomitant medication
Tender and swollen joints | Month 1, 3, 6, 9 and 12.
  Number of tender and swollen joints (range 0-30), higher values indicate more affected joints.
Physician-reported disease activity on a visual analogue scale | Month 1, 3, 6, 9 and 12.
  Patient-reported disease activity on a 0-100 mm scale; higher value indicate worse outcome.
Hand radiographs: Kellgren Lawrence | Month 6 and 12
  Conventional radiographs: change in radiographic severity according to Kellgren-Lawrence scale, range 0-4 in each joint higher value indicate worse outcome.
Hand radiographs: Verbruggen-Veys anatomical phase scoring system | Month 6 and 12
  Conventional radiographs: radiographic severity in finger joints according to Verbruggen-Veys anatomical phase scoring system, range 1-5; higher value indicate worse outcome.
Hand radiographs: OARSI atlas | Month 6 and 12
  Conventional radiographs: rdiographic severity according to the Osteoarthritis Research Society International (OARSI) atlas for the presence/severity of osteophytes, joint space narrowing and erosions.
Hand MRI | Month 6
  MRI of dominant hand: number of joints with synovitis and BMLs
Hand ultrasound | Month 1, 3, 6, 9 and 12.
  Ultrasound: number of finger joints with synovial thickening and power Doppler signals.
Knee ultrasound | Month 6
  Ultrasound: degree of synovitis in knee joints
Hip ultrasound | Month 6
  Ultrasound: degree of synovitis in hip joints
Adverse events | Through study completion, maximum 12 months, in addition to 3 months after end of treatment.
  Number of adverse events, serious adverse events, and withdrawals because of adverse events.

OTHER OUTCOMES:
Sub-study: biopsy of knee OA | Month 6
  Change in synovial cellular composition and gene expression with single-cell RNA sequencing analyses; subgroup analyses, n=16 patients
Sub-study: knee pain on a visual analogue scale | Month 6
  Self-reported knee pain previous 48 hours on a 0-100 mm scale at 6 months of treatment; higher value indicate worse outcome.
Question about blinding | Month 12
  The participants are asked which treatment they think they have received
HADS | Month 6
  Hospital Anxiety and Depression Scales (HADS), range 0-42, higher value indicate worse outcome.
PCS | Month 6
  Pain catastrophizing scale, range 0-12, higher value indicate worse outcome.
PSQ | Month 6
  Pain Sensitivity Questionnaire (PSQ), range 0-170, higher value indicate worse outcome.
Anchor questions for MCII and PASS | Month 6
  Questions about perceived improvement and acceptable symptom state that will be used to define minimally clinically important improvement and patient acceptable symptom state for other questionnaires
ASES | Month 6
  Arthritis Self Efficacy Scale (ASES), range 10-100, higher value indicate better outcome.
Pain sensitization | Month 6
  Pain sensitization: Pressure Pain Thresholds (PPT) by digital algometer; temporal summation by punctate probes; Conditioned Pain Modulation (CPM) by blood pressure ischemic test.
Soluble biomarkers of extracellular matrix turnover | Month 6 and 12
  Markers of collagen degradation (s-COMP, s-C1M, s-C2M, s-C3M, s-CTX1, sHA), collagen synthesis (s-proC2), aggrecan degradation (s-huARGS) and inflammation (s-calprotectin, s- vimentin, s-hsCRP and s-CRPM); Inflammatory cytokines (IL-1β, IL-1ra, IL-4, IL-6, IL-10, IL-12, IL-17, IL-18, IL-21, IFN-γ, TNF-α, VEGF, GM-CSF, CCL2, CCL3, CCL4, CXCL10) and hormones (leptin and resistin).
Omics | Month 6 and 12
  Omics analyses of whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, MD, PhD, Study Chair — Professor Em.
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
The trialists and other study personnel that conceive of the study, and then plan, manage, monitor, analyze and publish it, will have access to IPD. Participants' identification code numbers are de-identified by replacing the original code number with a new random code number. Only the PI and project coordinator have access to this code.
  The protocol, SAP, ICF, and CSR will be shared with regulatory agents as required.

REFERENCES:
- [Derived] Mathiessen A, Gaundal L, Sexton J, Sjolie D, Steen Pettersen P, Slatkowsky-Christensen B, Haugen IK. Protocol for the MERINO study: A randomized placebo-controlled trial assessing the efficacy, safety, and cost-effectiveness of methotrexate in people with erosive hand osteoarthritis. Osteoarthr Cartil Open. 2024 Dec 15;7(1):100558. doi: 10.1016/j.ocarto.2024.100558. eCollection 2025 Mar. PMID 39807424
- Available data/document: Study Protocol — https://drive.google.com/file/d/1AKuis2zJlqhUqY4OEPyVhQPpIiuPnnhr/view?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1mB2pEgRmuMhaVM_eNnnyXdqsyev4wev5/view?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1oE_9J-5uwLpboVWEsUJL6tHn4st1ea9r/view?usp=sharing